CLINICAL TRIAL: NCT01046838
Title: SIDAMI - Sildenafil and Diastolic Dysfunction After AMI
Brief Title: SIDAMI - Sildenafil and Diastolic Dysfunction After Acute Myocardial Infarction (AMI)
Acronym: SIDAMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jacob E Mueller (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Jacob E Mueller, MD, PhD, DmSci, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-011006-42
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Heart Failure, Diastolic
Keywords: Diastolic Heart Failure
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): placebo 3 x daily
  Interventions: Drug: Placebo
- sildenafil (Active Comparator): 40 mg sildenafil 3 x daily
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — 40 mg three times daily for 9 weeks
  Other Names: Revatio, Viagra
  Arms: sildenafil
Drug: Placebo — tablet 3 times daily for 9 weeks
  Arms: Placebo

SUMMARY:
In patients with Doppler echocardiographic signs of elevated LV filling pressures despite preserved LV systolic function after AMI treatment with the phosphodiesterase inhibitor sildenafil 40 mg three times daily for 9 weeks will compared with placebo

1. Improve resting LV filling and cardiac hemodynamics.
2. Improve exercise capacity.
3. Improve filling pattern and cardiac hemodynamics during exercise.

DETAILED DESCRIPTION:
Background:

Acute myocardial infarction (AMI) is characterized by regional myocardial damage which may lead to systolic and diastolic dysfunction with a subsequent risk of left ventricular (LV) remodeling, local and systemic neurohormonal activation, vascular dysfunction and development of heart failure. The pathophysiology and prognosis of LV systolic dysfunction after AMI has been the focus of research for several decades. Insights from these studies have led to several therapeutic interventions that improve outcome. In addition to depressed systolic function, clinical or radiographic evidence of heart failure is a consistent and powerful predictor of outcome in patients following AMI. Pulmonary congestion after AMI reflects raised LV filling pressures but is frequently seen after what appears to be only minor myocardial damage. The pathophysiological mechanism for this is incompletely understood but may involve impaired active relaxation of the myocardium and increased LV chamber stiffness, hence, abnormalities in diastolic function. Abnormal LV diastolic function especially when chamber stiffness is increased is characterized by a disproportionate increase in filling pressure during exercise and an inadequate increase of cardiac output. During ventricular diastole the left atrium acts as a conduit between the left ventricle and the pulmonary veins. Thus in case of increased filling pressures left atrial pressure is elevated exposing the pulmonary vascular bed to increased pressures. In accordance pulmonary artery pressure is frequently increased after AMI, even when systolic function is preserved.

Several recent studies have demonstrated that Doppler echocardiographic indices suggestive of increased filling pressure and increased pulmonary arterial pressure are associated with excess mortality and morbidity after AMI . The optimal management of this large group of patients is unknown, but in theory lowered preload improved cardiac output especially during exercise and lowering of pulmonary arterial pressure could relive symptoms and improve exercise capacity.

Sildenafil is a potent selective phosphodiesterase inhibitor that suppresses degradation of cyclic GMP. In the pulmonary bed this leads to pulmonary vasodilation, in addition sildenafil has been shown to improve endothelium dependent vasodilation thus augmenting abnormal vascular tone . In patients with systolic heart failure sildenafil has been demonstrated to lower pulmonary wedge pressure, improve cardiac index and lower pulmonary arterial pressure without causing systemic hypotension . Thus in theory sildenafil may have beneficial effects in patients at high risk of heart failure.

Hypothesis:

In patients with Doppler echocardiographic signs of elevated LV filling pressures despite preserved LV systolic function after AMI treatment with the phosphodiesterase inhibitor sildenafil 40 mg three times daily for 9 weeks will compared with placebo

1. Improve resting LV filling and cardiac hemodynamics.
2. Improve exercise capacity.
3. Improve filling pattern and cardiac hemodynamics during exercise.

Specific aims

Primary aims:

Among 70 patients with a recent AMI randomized to treatment with sildenafil 40 mg three times daily compared with placebo for 9 weeks to compare

1. mitral filling pattern, diastolic E/e´ ratio and left atrial volume,
2. pulmonary wedge pressure, cardiac index and pulmonary artery pressure, at rest and during submaximal exercise.

Secondary Aims Among 70 patients with a recent AMI randomized to sildenafil 40 mg three times daily compared with placebo to compared exercise capacity judged by bicycle ergometer testing.

Among 70 patients with a recent AMI randomized to sildenafil 40 mg three times daily compared with placebo to compared changes in NT-pro BNP.

Among 70 patients with a recent AMI randomized to sildenafil 40 mg three times daily compared with placebo to compared changes in diastolic E/e´ ratio during submaximal exercise.

Among 70 patients with a recent AMI randomized to sildenafil 40 mg three times daily compared with placebo to compare regional systolic function assessed with tissue tracking.

Tertiary aims

To assess the correlation between diastolic E/e' and Doppler assessed cardiac index during rest and exercise with pulmonary wedge pressure and cardiac index respectively.

To assess the association between exercise capacity and diastolic E/e', LA volume, and nt-proBNP.

Among 70 patients with a recent AMI randomized to sildenafil 40 mg three times daily compared with placebo to compare the prevalence of atrial arrhythmias after 9 weeks treatment.

Methods

Design The study is a prospective single center randomized double blind study. Eligible patients will be randomized to either conventional management and sildenafil for 4 months; or conventional management and placebo treatment.

Inclusion criteria

* Age >50 years
* Recent AMI (within 21 days) defined according to ESC/ACC guidelines
* Doppler echocardiographic signs of elevated filling pressures defined as

  * diastolic E/e' ratio >15, or
  * diastolic E/e' ratio 8-15 and left atrial volume index>32 ml/m2
* Preserved LV systolic function (EF>45%)
* Written informed consent

Exclusion criteria

* Ongoing myocardial ischemia
* Ongoing treatment with nitrates.
* Poor echocardiographic window
* Inability to exercise
* Permanent atrial fibrillation or paced rhythm
* Planned coronary artery bypass grafting
* Other noncardiac condition with expected survival less than 6 months
* Unwilling to participate
* Known intolerance to sildenafil

Study procedures

In possibly eligible patients a screening echocardiography is performed during hospitalization at the coronary care unit 2144 or 3141 HS Rigshospitalet, Denmark. If eligible and consent is obtained during hospitalisation an ambulatory exercise Doppler echocardiography with simultaneous invasive recording of pulmonary wedge pressure, pulmonary artery pressure and cardiac index and a 6 min walk test and maximal exercise test is performed 1 week after revascularization. Patients are then randomized in a 1 to 1 fashion to placebo or sildenafil 20 mg three times daily. If tolerated dosage is titrated every 2'nd week in the outpatient clinic to a target dose of 40 mg three times daily. After 9 weeks of treatment exercise echocardiography and 6 min walk test are repeated, in addition conventional maximal ergometer testing is performed.

Screening echocardiography 2 dimensional echocardiographic will be obtained from the parasternal and apical windows. Pulsed Doppler measurements of mitral inflow will be obtained with the transducer in the apical four-chamber view, with a 1-2 mm Doppler sample volume placed between the tips of mitral leaflets during diastole. Tissue Doppler imagining of the mitral annulus will be obtained from the apical 4-chamber view with a 1.5-mm sample volume placed at the medial mitral annulus. All Doppler echocardiographic examinations are done with horizontal sweep set to 100 mm/s. At least 3-5 cardiac cycles will be measured. LA volume will be obtained from the apical 4 and 2 chamber views with a zoomed image of the left atrium. Clinically indicted echocardiograms performed in the echolab may be used as screening echocardiograms.

* Wall motion index will semiquantitatively using a descending scoring as previously validated.
* Maximal left atrial volume will be measured at end-systole with the use of two orthogonal apical views.
* From the pulsed wave mitral inflow signal, peak E wave velocity will be measured.
* From the tissue Doppler assessment of the medial mitral annulus early (E') diastolic velocity will be recorded. Diastolic E/e' ratio will be calculated.

Resting echocardiography Doppler echocardiography will be performed on a GE medical Vivid 7 ultrasound machine by a single investigator. Images will be obtained from the parasternal and apical windows. M-mode recordings will be done in the parasternal long-axis view. Pulsed Doppler measurements of mitral inflow will be obtained with the transducer in the apical four-chamber view, with a 1-2 mm Doppler sample volume placed between the tips of mitral leaflets during diastole. Tissue Doppler imagining of the mitral annulus will be obtained from the apical 4-chamber view with a 1.5-mm sample volume placed at the medial and lateral mitral annulus. All Doppler echocardiographic examinations are done with horizontal sweep set to 100 mm/s. At least 3-5 cardiac cycles will be measured. Finally color coded real time tissue Doppler images will be acquired in the apical windows, with the lowest possible depth and smallest angle.

* End-systolic, end-diastolic volume and ejection fraction will be calculated according to the Simpson modified biplane method.
* Wall motion index will semiquantitatively be assessed according to the recommendations of the American Society of Echocardiography.
* Maximal left atrial volume will be measured at end-systole with the use of two orthogonal apical views with zoom of the left atrium.
* From the pulsed wave mitral inflow signal, peak E wave velocity, peak A wave velocity, and mitral E-wave deceleration time will be measured.
* From peak tricuspid regurgitant velocity and size of inferior v. cava pulmonary arterial systolic pressure will be estimated.
* From the tissue Doppler assessment of the medial mitral annulus early (E') diastolic velocity will be recorded. Diastolic E/e' ratio will be calculated.
* From color coded tissue Doppler images systolic longitudinal fibre shortening will be assessed using tissue tracking.
* From 2dimensional images speckle tracing will be performed to assess radial and longitudinal LV function.

Exercise echocardiography Exercise echocardiography is performed at cardiac intensive care unit 2143. Before exercise a Swan Ganz catheter is introduced with a seldinger technique through the right jugular vein. Simultaneous with resting echocardiography pulmonary artery pressure, left atrial pressure, cardiac index and pulmonary wedge pressure is recorded. Patients are then exercised on a supine bicycle with increasing workload to 100W with increments of 25W every 2'nd min. At 100W echocardiography is repeated with simultaneous assessment of pulmonary artery pressure, left atrial pressure, pulmonary wedge pressure and cardiac index.

Neurohormonal analyses Prior to surgery and at each follow-up visit venous blood samples will be drawn for analysis of plasma N-terminal proBNP, and of plasma N-terminal ANP concentrations. In addition plasma will be frozen at each visit for possible later analysis.

Six minutes walk test A 6 min. walk test will be performed at baseline 9 weeks.

Exercise test A conventional bicycle ergometer test is performed at hospital discharge and after 4 months. Maximal exercise is achieved by increments on 25W every 2'nd min. with continuous ECG recording and assessment of blood pressure every 2'nd min.

Feasibility and sample size estimation From a recent study at a tertiary invasive centre including 380 patients with AMI, (Aberdeen AMI study, Hillis et al ESC 2006), it was found that among 219 patients EF was >45%. Among those patients E/e' >15 was found in 41 patients, and in further 48 E/e' 8-15 and left atrial volume index >32 ml/m2 was found. Thus 40% of patients with LVEF>45% would be potentially eligible. Annually 2500 patients are admitted or transferred to RH with AMI.

Based on a standard deviation of E/e' of 5 (estimated from potentially eligible patients from the Aberdeen AMI study), an alpha of 0.05 and beta of 0.80 a sample of 70 patients will allow detection of a difference in E/e' of 3.6. Sample size estimation is performed according to Altmann using nomogram.

ELIGIBILITY:
Inclusion Criteria:

* Age >50 years
* Recent AMI (within 21 days) defined according to ESC/ACC guidelines
* Doppler echocardiographic signs of elevated filling pressures defined as

  * diastolic E/e' ratio >15, or
  * diastolic E/e' ratio 8-15 and left atrial volume index>32 ml/m2
* Preserved LV systolic function (EF>45%)
* Written informed consent

Exclusion Criteria:

* Ongoing myocardial ischemia
* Ongoing treatment with nitrates.
* Poor echocardiographic window
* Inability to exercise
* Permanent atrial fibrillation or paced rhythm
* Planned coronary artery bypass grafting
* Other noncardiac condition with expected survival less than 6 months
* Unwilling to participate
* Known intolerance to sildenafil
* Non-arteritic anterior ischaemic optic neuropathy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-12; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Among 70 patients with a recent AMI randomized to sildenafil 40 mg three times daily compared with placebo to compared Pulmonary wedge pressure, cardiac index and pulmonary artery pressure, at rest and during submaximal exercise. | 9 weeks

SECONDARY OUTCOMES:
Among 70 patients with a recent AMI randomized to sildenafil 40 mg three times daily compared with placebo to compared exercise capacity judged by bicycle ergometer testing. | 9 weeks
Among 70 patients with a recent AMI randomized to sildenafil 40 mg three times daily compared with placebo to compared changes in NT-pro BNP. | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jacob E Møller, MD, Phd, DmSci, Principal Investigator — Rigshospitalet, Denmark; Mads J Andersen, MD, Principal Investigator — The Heart Center, Cardiology
Locations (1):
- Rigshospitalet, Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Andersen MJ, Wolsk E, Bakkestrom R, Christensen N, Carter-Storch R, Omar M, Dahl JS, Frederiksen PH, Borlaug B, Gustafsson F, Hassager C, Moller JE. Pressure-flow responses to exercise in aortic stenosis, mitral regurgitation and diastolic dysfunction. Heart. 2022 Nov 10;108(23):1895-1903. doi: 10.1136/heartjnl-2022-321204. PMID 36356959
- [Derived] Andersen MJ, Ersboll M, Axelsson A, Gustafsson F, Hassager C, Kober L, Borlaug BA, Boesgaard S, Skovgaard LT, Moller JE. Sildenafil and diastolic dysfunction after acute myocardial infarction in patients with preserved ejection fraction: the Sildenafil and Diastolic Dysfunction After Acute Myocardial Infarction (SIDAMI) trial. Circulation. 2013 Mar 19;127(11):1200-8. doi: 10.1161/CIRCULATIONAHA.112.000056. Epub 2013 Feb 13. PMID 23406672